CLINICAL TRIAL: NCT04648033
Title: A Phase I Trial of the Hypoxia Modifier Atovaquone in Combination With Radical Concurrent Chemoradiotherapy in Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Atovaquone With Radical ChemorADIotherapy in Locally Advanced NSCLC
Acronym: ARCADIAN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Cancer Research UK (Other); National Institute for Health Research, United Kingdom (Other Government); NHS Lothian (Other Government); Oxford University Hospitals NHS Trust (Other); NHS Research Scotland (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_088
Record Dates: First submitted 2020-10-08; First posted 2020-12-01 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2023-05

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer
MeSH Terms: interventions — Atovaquone; Cisplatin; Vinorelbine

STUDY DESIGN:
Intervention Model Description: Time-to-Event Continual Reassessment Method to determine the maximum tolerated dose (MTD) of atovaquone in combination with concurrent CRT in NSCLC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose level 1 - 450 mg BD atovaquone + concurrent CRT (Experimental): Atovaquone:
  * Taken during an initial run in period (2 weeks +/- 7 days), then continued during standard of care chemoradiotherapy.
  * One of 4 dose levels is allocated to each patient by a TiTE-CRM statistical model which takes into account all toxicity data to date.
  * Dose levels - 450 mg, 600 mg, 675 mg or 750 mg (all doses PO BD).
  * Last dose atovaquone taken on the last day of radiotherapy.
  * Total duration of atovaquone treatment is 59 days (+/- 7 days), unless stopped earlier for toxicity or any other reason.
  Chemotherapy:
  * 2 x 21-day cycles.
  * 80 mg/m2 cisplatin on day 1 and 22 of chemoradiotherapy.
  * 15 mg/m2 vinorelbine on days 1,8, 22 and 29 of chemoradiotherapy.
  Radiotherapy:
  * 66 Gy in 33 fractions.
  * Delivered once daily, 5 days a week (Monday-Friday) for 6.5 weeks.
  Interventions: Drug: Atovaquone Oral Suspension; Drug: Standard of care chemotherapy; Radiation: Standard of care radiotherapy
- Dose level 2 - 600 mg BD atovaquone + concurrent CRT (Experimental): Atovaquone:
  * Taken during an initial run in period (2 weeks +/- 7 days), then continued during standard of care chemoradiotherapy.
  * One of 4 dose levels is allocated to each patient by a TiTE-CRM statistical model which takes into account all toxicity data to date.
  * Dose levels - 450 mg, 600 mg, 675 mg or 750 mg (all doses PO BD).
  * Last dose atovaquone taken on the last day of radiotherapy.
  * Total duration of atovaquone treatment is 59 days (+/- 7 days), unless stopped earlier for toxicity or any other reason.
  Chemotherapy:
  * 2 x 21-day cycles.
  * 80 mg/m2 cisplatin on day 1 and 22 of chemoradiotherapy.
  * 15 mg/m2 vinorelbine on days 1,8, 22 and 29 of chemoradiotherapy.
  Radiotherapy:
  * 66 Gy in 33 fractions.
  * Delivered once daily, 5 days a week (Monday-Friday) for 6.5 weeks.
  Interventions: Drug: Atovaquone Oral Suspension; Drug: Standard of care chemotherapy; Radiation: Standard of care radiotherapy
- Dose level 3 - 675 mg BD atovaquone + concurrent CRT (Experimental): Atovaquone:
  * Taken during an initial run in period (2 weeks +/- 7 days), then continued during standard of care chemoradiotherapy.
  * One of 4 dose levels is allocated to each patient by a TiTE-CRM statistical model which takes into account all toxicity data to date.
  * Dose levels - 450 mg, 600 mg, 675 mg or 750 mg (all doses PO BD).
  * Last dose atovaquone taken on the last day of radiotherapy.
  * Total duration of atovaquone treatment is 59 days (+/- 7 days), unless stopped earlier for toxicity or any other reason.
  Chemotherapy:
  * 2 x 21-day cycles.
  * 80 mg/m2 cisplatin on day 1 and 22 of chemoradiotherapy.
  * 15 mg/m2 vinorelbine on days 1,8, 22 and 29 of chemoradiotherapy.
  Radiotherapy:
  * 66 Gy in 33 fractions.
  * Delivered once daily, 5 days a week (Monday-Friday) for 6.5 weeks.
  Interventions: Drug: Atovaquone Oral Suspension; Drug: Standard of care chemotherapy; Radiation: Standard of care radiotherapy
- Dose level 4 - 750 mg BD atovaquone + concurrent CRT (Experimental): Atovaquone:
  * Taken during an initial run in period (2 weeks +/- 7 days), then continued during standard of care chemoradiotherapy.
  * One of 4 dose levels is allocated to each patient by a TiTE-CRM statistical model which takes into account all toxicity data to date.
  * Dose levels - 450 mg, 600 mg, 675 mg or 750 mg (all doses PO BD).
  * Last dose atovaquone taken on the last day of radiotherapy.
  * Total duration of atovaquone treatment is 59 days (+/- 7 days), unless stopped earlier for toxicity or any other reason.
  Chemotherapy:
  * 2 x 21-day cycles.
  * 80 mg/m2 cisplatin on day 1 and 22 of chemoradiotherapy.
  * 15 mg/m2 vinorelbine on days 1,8, 22 and 29 of chemoradiotherapy.
  Radiotherapy:
  * 66 Gy in 33 fractions.
  * Delivered once daily, 5 days a week (Monday-Friday) for 6.5 weeks.
  Interventions: Drug: Atovaquone Oral Suspension; Drug: Standard of care chemotherapy; Radiation: Standard of care radiotherapy

INTERVENTIONS:
Drug: Atovaquone Oral Suspension — Atovaquone, cisplatin and vinorelbine are all considered Investigational Medicinal Products (IMPs) in this trial due to the investigation of these drugs in a novel combination. Patients will be allocated one of four doses of atovaquone: 450 mg, 600 mg, 675 mg or 750 mg (all doses PO BD).
  Other Names: Wellvone
Drug: Standard of care chemotherapy — Atovaquone, cisplatin and vinorelbine are all considered Investigational Medicinal Products (IMPs) in this trial due to the investigation of these drugs in a novel combination. Patients will receive two 21-day cycles of cisplatin and vinorelbine chemotherapy, comprising 80 mg/m2 cisplatin on days 1 & 22 of their CRT treatment and 15 mg/m2 vinorelbine on days 1, 8, 22 & 29.
  Other Names: Cisplatin; Vinorelbine
Radiation: Standard of care radiotherapy — Thoracic radiotherapy will commence on day one of chemotherapy and be delivered in 66 Gy in 33 fractions, once daily, 5 days a week (Monday-Friday) for 6.5 weeks.

SUMMARY:
This is a phase I, open-label trial that will utilise a Time To Event Continual Reassessment Method (TiTE-CRM) to determine the maximum tolerated dose (MTD) of atovaquone in combination with concurrent CRT in NSCLC. Twenty evaluable participants will be recruited at three centres.

DETAILED DESCRIPTION:
Twice daily oral atovaquone will be added to standard concurrent chemoradiotherapy (CRT): 66 Gy in 33 fractions, once daily, 5 days a week (Monday-Friday), with cisplatin (80 mg/m2 IV on days 1 and 22 of CRT) and vinorelbine (15 mg/m2 IV on days 1, 8, 22 and 29 of CRT). Whilst awaiting CRT to start, patients will receive two weeks (+/- 7 days) of oral atovaquone to ensure steady state is reached (after seven days). Patients will be allocated one of four dose levels: 450 mg, 600 mg, 675 mg or 750 mg (all doses PO BD). Atovaquone dose will be assigned as per the TiTE-CRM statistical model. The first two trial participants will receive 450 mg BD. In the absence of unacceptable toxicity, subsequent patients will be assigned doses up to and including 750 mg BD.

Hypoxia biomarker data will be collected at baseline (start of atovaquone run-in) and following two weeks (+/- 7 days) of atovaquone treatment. Atovaquone will then be continued without break for the duration of CRT, with the CRT schedule remaining constant for all patients at both centres. Assessment for Dose Limiting Toxicities (DLTs) will be from the first scheduled dose of atovaquone until three months after completion of CRT. The CT scan performed at the three-month follow up visit will be reviewed to collect tumour response data.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for inclusion in this study if all of the following criteria apply:

1. Histologically or cytologically confirmed diagnosis of locally advanced NSCLC and selected for treatment with full dose radical concurrent CRT
2. At least one measurable lesion greater than 2 cm maximal length in any direction on routine imaging (CT or PET-CT scan performed in the 60 days prior to consent)
3. Male or female, age at least 18 years
4. ECOG performance status 0 or 1
5. Adequate pulmonary function tests for thoracic radiotherapy (FEV1 and TLCO, greater than 40 percent predicted)
6. Haematological and biochemical indices within the ranges shown below:

   Bilirubin ≤ 1.5 x upper limit of normal (ULN); ALT and/or AST ≤ 2.5 x ULN; Creatinine clearance ≥ 60 mL/min; Absolute Neutrophil Count ≥ 1.5 x 10*9/L; Platelets ≥ 100 x 10*9/L; Haemoglobin ≥ 90 g/L; INR ≤ 1.5
7. The patient is willing and able to comply with the protocol scheduled follow-up visits and examinations for the duration of the study
8. Written (signed and dated) informed consent and be capable of co-operating with protocol

Exclusion Criteria:

1. Pregnant or breast-feeding women, or women of childbearing potential unless effective methods of contraception are used
2. Previous systemic chemotherapy or biological therapy within 21 days of commencing atovaquone treatment
3. Treatment with any other investigational agent as part of a clinical trial within 28 days of study enrolment
4. Previous thoracic radiotherapy
5. Known previous adverse reaction to atovaquone or its excipients
6. Active hepatitis, gallbladder disease or pancreatitis
7. Impaired gastrointestinal function that may significantly alter absorption of atovaquone
8. Concurrent administration of warfarin in the 14 days prior to starting atovaquone
9. Concurrent administration of known electron transport chain inhibitors (e.g. metformin). A wash-out period prior to administration of atovaquone is required (e.g. 4 days for metformin).
10. An additional cancer diagnosis that the treating clinician feels may significantly impact planned CRT treatment tolerability or treatment outcome
11. Established diagnosis of pulmonary fibrosis
12. Established diagnosis of connective tissue disorder (e.g. scleroderma or systemic lupus erythematosus)
13. Cardiac morbidity such as angina, myocardial infarction in the previous six months, unstable angina or uncontrolled hypertension, left ventricular failure or severe valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Higgins, Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - Western General Hospital, NHS Lothian, Edinburgh
  - Guy's and St Thomas', London
  - Churchill Hospital, Oxford University Hospitals, Oxford

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Started | 3 | 2 | 1 | 15
Completed | 3 | 2 | 1 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT | Total
Number analyzed (Participants) | 3 | 2 | 1 | 15 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (17.7) | 48.0 (9.9) | 65.0 (NA) — Only 1 participant was registered to this group. | 65.2 (16.4) | 63.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 6 | 7
  Male | 3 | 1 | 1 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 1 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 6 | 6
Smoking status [Count of Participants; unit: Participants]
  Never smoked | 1 | 1 | 0 | 0 | 2
  Ex-smoker | 2 | 0 | 1 | 13 | 16
  Current smoker | 0 | 1 | 0 | 2 | 3
Non-small cell lung cancer sub-type [Count of Participants; unit: Participants]
  Adenocarcinoma | 3 | 1 | 0 | 4 | 8
  Squamous cell carcinoma | 0 | 1 | 1 | 11 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities in Patients Taking Atovaquone in Combination With Radical Concurrent Chemoradiotherapy for Non-small Cell Lung Cancer.
Description: To determine the maximum tolerated dose level (and therefore recommended phase II dose) of atovaquone when administered concomitantly with radical concurrent chemoradiotherapy (CRT) in patients with non-small cell lung cancer (NSCLC). This is the dose of atovaquone associated with no more than 48% dose limiting toxicity (DLT) rate (target toxicity level).
Time Frame: From first dose of atovaquone to 3-month follow up visit (up to 25 weeks)
Measure: Number; unit: Dose Limiting Toxicities (DLTs)
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 3 | 2 | 1 | 15
Dose Limiting Toxicities (DLTs) | 0 | 0 | 0 | 2
Statistical Analysis 1: Comparison: Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT vs Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT vs Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT vs Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT; The primary analysis is performed using the Time-To-Event Continual Reassessment Method (TiTE-CRM). Giving posterior estimates for the probability of toxicity (DLT) at each dose level; Test type: Other; Probability of DLT at dose level 4 = 0.116, 95% CI 2-sided [0.032 to 0.26]

2. Secondary Outcome: Severity of Worst Adverse Events Per Dose Level of Atovaquone Administered in Combination With Radical Concurrent Chemotherapy for NSCLC According to CTCAE V4.03
Description: Toxicity profile when atovaquone administered in combination with radical concurrent chemotherapy for NSCLC. Worst grade adverse event for each patient by dose schedule (according to the Common Terminology Criteria for Adverse Events, Version 4.03). Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe or medically significant, but not immediately life-threatening); Grade 4 (life-threatening); Grade 5 (death).
Time Frame: From first dose of atovaquone until last follow up visit at 6 months post completion of CRT (up to 38 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 3 | 2 | 1 | 15
Participants
  Worst AE: Grade 1 | 0 | 0 | 1 | 0
  Worst AE: Grade 2 | 1 | 1 | 0 | 6
  Worst AE: Grade 3 | 2 | 1 | 0 | 6
  Worst AE: Grade 4 | 0 | 0 | 0 | 1
  Worst AE: Grade 5 | 0 | 0 | 0 | 2

3. Secondary Outcome: Number of Patients for Whom it Was Possible to Derive a Hypoxia Metagene Signature Score From 3'RNA-Seq of Genetic Material From Archival Tumour Samples
Description: To confirm feasibility of measuring hypoxia metagene signature using 3'RNA-Seq on genetic material extracted from diagnostic non-small cell lung tumour samples. The score method was derived by Buffa et al (Buffa et al. Large meta-analysis of multiple cancers reveals a common, compact and highly prognostic hypoxia metagene. Br J Cancer. 2010 Jan 19;102(2):428-35. doi: 10.1038/sj.bjc.6605450).
Time Frame: At baseline (diagnosis)
Population: Five of 21 participants did not have a hypoxia metagene signature score derived due to the quality of extracted RNA being of insufficient quality to sequence (n=3), no archival tumour sample being available (n=1), or participant withdrew consent (n=1).
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 3 | 2 | 0 | 11
Participants | 3 | 2 | 0 | 11

4. Secondary Outcome: Mean Baseline Tumour Hypoxia Level (TBRvol) Assessed by F18-FMISO PET-CT
Description: The level of hypoxia in patient tumours was calculated using the Tumour-to-Blood Ratio volume (TBRvol) assessed from the patient's baseline PET scan. This scan was conducted with 18F-labelled fluoromisonidazole (F18-FMISO) which has been shown to selectively bind to hypoxic cells and can be quantified with PET imaging (Koh, et al. Imaging of hypoxia in human tumours with [F-18]fluoromisonidazole. Int J Radiat Oncol Biol Phys. 1992;22(1)). Tumour outlining of the region of interest on each axial slice was conducted centrally for all patients in consultation with an experienced consultant radiologist and combined to give a volume of interest (VOI). The number of voxels in the VOI with a threshold regional tumor:plasma F18-FMISO ratio of greater than or equal to 1.4 were combined to give the TBRvol (above reference). Patients with a TBRvol at baseline of <1.5mL were regarded as unevaluable for later endpoints, so are excluded from the report.
Time Frame: At baseline (prior to atovaquone treatment)
Population: Nine of 21 patients results were excluded from the report because they did not have F18-FMISO PET-CT scans at two of two timepoints in the trial (e.g. due to having a TBRvol considered too low to be evaluable on the first scan (n=6), or for logistical reasons (n=3)).
Measure: Mean (Full Range); unit: TBRvol (mL)
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 2 | 1 | 0 | 9
TBRvol (mL) | 282.4 [4.4 to 560.4] | 21.4 [NA to NA] — There was only one participant in this group (for reasons given in analysis population description, above), so range is not applicable. |  | 58.7 [2.6 to 162.0]

5. Secondary Outcome: Mean Baseline Plasma miR-210 Level Assessed Via TaqMan Quantitative PCR
Description: MicroRNA-210 (miR-210) has been found to be upregulated in response to hypoxia-inducing factors (Dang and Myers, The Role of Hypoxia-Induced miR-210 in Cancer Progression, Int. J. Mol. Sci., vol 16, 2015). Additionally, elevated serum levels of miR-210 are indicative of poor clinical outcomes in non-small cell lung cancer (He, et al. Clinical Significance of miR-210 and its Prospective Signaling Pathways in Non-Small Cell Lung Cancer. Physiol. Biochem. Int. J. Exp. Cell. Physiol. Biochem. Pharmacol., vol. 46, 2018). RNA was isolated from blood plasma and miR210 level detected using a two-step TaqMan quantitative PCR, using TaqMan probes for miR-210. An endogenous control miRNA (miR-16), plus an exogenous synthetic miRNA (cel-miR-39) were used for normalisation of miR210 counts. This endpoint was assessed in order to investigate a possible alternative to 18F-FMISO PET-CT scan for assessment of patients' tumour hypoxia level.
Time Frame: At baseline (prior to atovaquone treatment)
Population: Eight of 21 participant samples are not reported either because the samples showed evidence of haemolysis (n=7) or because the participant withdrew consent (n=1).
Measure: Mean (Full Range); unit: miR210 count (x10^3)
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 2 | 1 | 0 | 10
miR210 count (x10^3) | 0.00146 [0.00142 to 0.00149] | 0.00219 [NA to NA] — There was only one participant analysed this group (for reasons given in analysis population description, above), so range is not applicable. |  | 0.00195 [0.00098 to 0.00451]

6. Secondary Outcome: Mean Percentage Change in Tumour Hypoxia Level Between Baseline and After Two Weeks (+/- 7 Days) of Atovaquone Treatment
Description: The level of hypoxia (Tumour-to-Blood Ratio volume, TBRvol) in patient tumours was calculated at baseline and following two weeks (+/- 7 days) of atovaquone treatment according to the details given in outcome measure 4. The mean percentage difference in TBRvol between the two timepoints at each dose level of atovaquone was calculated and is reported, below. Patients with a TBRvol at baseline of <1.5mL were regarded as unevaluable as it would not be possible to evaluate a reduction in hypoxic volume between this timepoint and the later timepoint. These patients were excluded from the report.
Time Frame: Between baseline (prior to atovaquone treatment) and following two weeks (+/- 7 days) of atovaquone treatment (up to 21 days)
Population: as for outcome 4
Measure: Mean (Full Range); unit: Percentage change in TBRvol
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 2 | 1 | 0 | 9
Percentage change in TBRvol | -8 [-37 to 22] | -15 [NA to NA] — There was only one participant analysed in this group (see analysis population description, above), therefore range is not applicable. |  | -25 [-91 to 4]

7. Secondary Outcome: Mean Percentage Change in Plasma miR-210 Level Between Baseline and After Two Weeks (+/- 7 Days) of Atovaquone Treatment, Assessed Via TaqMan Quantitative PCR
Description: The miR-210 in participant plasma samples was calculated at baseline and following two weeks (+/- 7 days) of atovaquone treatment according to the details given in outcome measure 5. The mean percentage difference in miR210 count between the two timepoints for each dose level of atovaquone was calculated and is reported, below. This endpoint was assessed in order to investigate a possible alternative to 18F-FMISO PET-CT scan for assessment of patients' tumour hypoxia level.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Mean (Full Range); unit: Percentage change in miR210 count
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 2 | 1 | 0 | 10
Percentage change in miR210 count | 53.0 [50.9 to 55.1] | -42.5 [NA to NA] — There was only one participant analysed this group (for reasons given in analysis population description, above), so range is not applicable. |  | 15.1 [-33.0 to 91.7]

8. Secondary Outcome: Objective Tumour Response to Treatment With Atovaquone in Combination With Chemoradiotherapy, as Evaluated by CT or PET-CT Scan and Quantified by RECIST 1.1
Description: Efficacy of the combination (atovaquone and chemoradiotherapy), measured by objective tumour response via RECIST 1.1 (Eisenhauer, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45(2):228-247). Scale of response assessed as Progressive Disease (PD) (worst outcome), Stable Disease (SD), Partial Response (PR), Complete Response (CR) (best outcome).
Time Frame: At 3 months post completion of chemoradiotherapy (up to 25 weeks after first dose of atovaquone)
Population: Two of 21 participants were non-evaluable because they did not have a follow up scan at 3 months post-chemoradiotherapy treatment on which RECIST assessment could be performed. .
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
Number analyzed (Participants) | 3 | 2 | 1 | 13
Participants
  Complete Response (CR) | 0 | 0 | 0 | 1
  Partial Response (PR) | 2 | 2 | 1 | 7
  Stable Disease (SD) | 1 | 0 | 0 | 2
  Progressive Disease (PD) | 0 | 0 | 0 | 3

ADVERSE EVENTS:
Time Frame: Adverse events (including serious events) are reported from first dose of atovaquone to last follow up visit at 6 months post chemoradiotherapy (up to 38 weeks).
Arm/Group | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/1 | 2/15
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/2 | 0/1 | 7/15
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 1/1 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT (N=3) | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT (N=2) | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT (N=1) | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT (N=15)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 450 mg BD Atovaquone + Concurrent CRT (N=3) | Dose Level 2 - 600 mg BD Atovaquone + Concurrent CRT (N=2) | Dose Level 3 - 675 mg BD Atovaquone + Concurrent CRT (N=1) | Dose Level 4 - 750 mg BD Atovaquone + Concurrent CRT (N=15)
Blood & Lymphatic System Disorders (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 0 (0) | 3 (8)
Cardiac Disorders (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorders (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye disorders (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 3 (5) | 2 (16) | 1 (3) | 14 (45)
General Disorders & Administration Site Conditions (General disorders) | 3 (3) | 2 (3) | 1 (1) | 11 (22)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections & Infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Investigations (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Metabolism & Nutrition Disorders (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 8 (16)
Musculoskeletal & Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (4)
Nervous System Disorders (Nervous system disorders) | 2 (5) | 1 (1) | 0 (0) | 9 (15)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8)
Renal and urinary disorders (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 11 (27)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 4 (5)
Vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT04648033/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT04648033/SAP_001.pdf